CLINICAL TRIAL: NCT00970476
Title: Response To Cardiac Resynchronization Therapy In Heart Failure: Role Of Arterial Stiffness
Status: Withdrawn | Type: Observational
Why Stopped: limited enrollment
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Other Study IDs: 06-14344
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Arterial Stiffness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine if arterial stiffness as measured by non-invasive pulse wave velocity can predict the response to resynchronization therapy in heart failure.

DETAILED DESCRIPTION:
The patients receiving CRT are medically refractory, symptomatic, NYHA class III or IV disease and QRS duration of 130 m sec or greater, and a left ventricular ejection fraction of 30 percent or less.

The pulse wave velocity between carotid and femoral (PWVcf) will be recorded in each subject at base line (before and after CRT), at one month (after AV delay optimization) and again at 6 months after CRT. The arterial pulse wave is recorded at a proximal artery, such as the carotid artery, and as well as at a distal artery, such as the femoral artery. The superficial location of the carotid and femoral arteries means that their pulse waveforms are readily measured noninvasively using the M Hz Doppler probe, and between these two sites the pulse wave has to travel through most of the aorta. The time delay between the arrival of a predefined part of the pulse wave, such as the foot, at these 2 points is obtained by gating to the peak of the R-wave of the ECG. The distance traveled by the pulse wave is measured over the body surface and PWV is then calculated as distance/time (m/s).

Clinical evidence of response: Either one or more of the following: 1) Improvement in NYHA functional classification, 2) Improvement in 6 minute walking distance. 3) Change in functional class, exercise tolerance while the heart is getting smaller on CXR. 4) Stabilization of patient CHF even without subjective improvement over 6 months (remaining class III rather than progressive to class IV). Imaging evidence of response: 1) Increase in left ventricular ejection fraction. 2) Reduction of mitral regurgitation. 3) Reduction of LV volume signifying reverse remodeling.

ELIGIBILITY:
Inclusion Criteria:

* The patients receiving CRT are medically refractory, symptomatic, NYHA class III or IV disease and QRS duration of 130 m sec or greater, and a left ventricular ejection fraction of 30 percent or less.
* All individuals are carefully selected after appropriate clinical evaluation as determined by the treating physicians to exclude possible reversible causes of heart failure.

Exclusion Criteria:

* Patients with permanent atrial fibrillation and non-palpable carotid and/or femoral pulses will be excluded due to technical limitations of the procedure used for the measurement of arterial stiffness.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients, who are scheduled to undergo cardiac resynchronization therapy (CRT) at Creighton University Cardiac Center will be included in this study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
If arterial stiffness can predict the response to resynchronization therapy in heart failure. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Siva Sontineni, M.D., Principal Investigator — Creighton Cardiac Center